CLINICAL TRIAL: NCT06556797
Title: How to Differentiate Congestive and Non-congestive Dyspnea in the Emergency Department? Proof-of-concept Study on Microperfusion Analysis Via GapCO2
Brief Title: Proof-of-concept Study on Dyspnea Analysis Via GapCO2
Acronym: MicroDys
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP221251; 2022-A01957-36 (Other: IDRCB ANSM)
Record Dates: First submitted 2024-06-21; First posted 2024-08-16 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Acute Dyspnea; Dyspnea
Keywords: Acute dyspnea; Emergency department; Dyspnea; Congestion; Proof-of-concept study; GapCO2
MeSH Terms: conditions — Dyspnea; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients presenting to the emergency department with acute dyspnea undergo arterial blood gas measurement and monitoring of transcutaneous capnography using the TCM5 monitor. The aim of this study is to determine whether GapCO2, the difference between transcutaneous and arterial pCO2 (PaCO2 - PtcCO2), is correlated with the congestive or non-congestive origin of dyspnea.

DETAILED DESCRIPTION:
Upon arrival at the emergency department, patients are placed in the vital emergency reception area for monitoring. An emergency physician will review the selection criteria and offer the patient participation. The information sheet will be provided to the patient along with a copy of the non-opposition form in case of patient agreement.

Before the introduction of any treatment, a TC 92 sensor is placed on the earlobe (or on the forehead if the earlobe is inaccessible), connected to a Radiometer TCM5 monitor, measuring SpO2 (Massimo technology), perfusion index, and transcutaneous capnography (PtcCO2).

After a 5-minute equilibration period, measurements were taken throughout the duration of patient management. Standard diagnostic and therapeutic management will be provided according to the attending physician's prescription. The attending physician won't consider PtcCO2 (nor GapCO2) measurements in patient management.

At the time of data analysis, an adjudication committee comprising 2 emergency physicians from the inclusion service but not involved in patient care will review the complete medical records of patients to determine whether dyspnea was of congestive or non-congestive origin.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patient presenting with acute dyspnea defined by a sensation of respiratory discomfort with at least one of the following criteria: RR ≥ 22 and/or SpO2 < 95%
* Arterial blood gas sampling performed as part of care
* Inclusion less than 1 hour after arrival time to the emergency department
* Non-opposition to participation in the study

Exclusion Criteria:

* Temperature greater than or equal to 37.5°C
* Patient who has already received a diuretic or vasodilator treatment in the emergency department or by a prehospital medical team
* Systolic blood pressure less than or equal to 100 mmHg and/or signs of peripheral hypoperfusion
* Inability to express refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient presenting to the emergency department of the inclusion center for acute dyspea
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2025-01-26 (Actual); Primary Completion 2026-03-26 (Estimated); Study Completion 2026-04-26 (Estimated)

PRIMARY OUTCOMES:
GapCO2 | Within 1 hour after enrolment
  PaCO2 measured via arterial blood gas analysis - PtcCO2 measured via TCM5 monitor, at 37°C

SECONDARY OUTCOMES:
Diagnostic performance of GapCO2 at 37°C | Within 1 hour after enrolment
Proportion of patients who underwent GapCO2 measurement among those who presented to the emergency department for dyspnea on the days of inclusion | up to 28 days
  Feasibility of measuring GapCO2 in the emergency department

CONTACTS AND LOCATIONS:
Overall Officials: Judith GORLICKI, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Emergency Department Hospital Avicenne, Bobigny, France

IPD SHARING:
Plan to Share IPD: No